CLINICAL TRIAL: NCT03164746
Title: Demonstration of the Effectiveness of Treatment by Therapeutic Body Wraps in Children and Adolescents Suffering From Autism Spectrum Disorder With Severe Injurious Behavior.
Brief Title: Treatment by Therapeutic Body Wraps in Children and Adolescents Suffering From Autism With Severe Injurious Behavior.
Acronym: PACKING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2007/0715; 2007-A01376-47 (Other: ID-RCB number, ANSM); DGS 2008-0070 (Other: DGS number)
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Therapeutic body wraps
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DRY group (Active Comparator): Dry sheet therapeutic body wraps will be conducted through twice-a-week sessions for a 3-month duration. Sessions take place in the same quiet room and they usually last 45 minutes each up to 1 hour depending on the patient's response. During sessions, the patient wearied a bathing suit. Sessions were conducted under the supervision of an occupational therapist and involved at least two members of the patient's care team.
  Interventions: Other: Dry sheet Therapeutic body wraps
- WET Group (Experimental): Wet sheet therapeutic body wraps will be conducted through twice-a-week sessions for a 3-month duration. Sessions take place in the same quiet room and they usually last 45 minutes each up to 1 hour depending on the patient's response. During sessions, the patient wearied a bathing suit. Sessions were conducted under the supervision of an occupational therapist and involved at least two members of the patient's care team.
  Interventions: Other: WET sheet Therapeutic body wraps

INTERVENTIONS:
Other: Dry sheet Therapeutic body wraps — At the beginning of the session, the patient's consent to proceed was orally obtained, as no session was compulsory. The therapists checked behavioral manifestations of refusal. Then, the patient was first wrapped in Dry damp sheets (cold phase) and covered up with a rescue and a dry blanket. Afterward the body spontaneously warmed up (warm phase). The patient was then invited to freely express his feelings.
  Arms: DRY group
Other: WET sheet Therapeutic body wraps — At the beginning of the session, the patient's consent to proceed was orally obtained, as no session was compulsory. The therapists checked behavioral manifestations of refusal. Then, the patient was first wrapped in wet damp sheets (cold phase) and covered up with a rescue and a dry blanket. Afterward the body spontaneously warmed up (warm phase). The patient was then invited to freely express his feelings.
  Arms: WET Group

SUMMARY:
Severe injurious behaviors in children with autism spectrum disorder are challenging. First line treatment approaches include behavioral techniques but pharmacotherapy is frequently required despite frequent adverse effects in youths.

Therapeutic body wraps has been reported in small series or case reports, but has never been assessed in the context of a randomized controlled trial.

The present study is an exploratory, multicenter, randomized, controlled, open label with blinded outcome assessment (PROBE design) trial of the effect of wet versus dry therapeutic body wraps in children presenting with autism spectrum disorder and severe injurious behavior.

DETAILED DESCRIPTION:
Packing therapy has never been assessed, namely in children with severe injurious behavior and autism spectrum disorder.

The aim of the present study is to evaluate the beneficial effect of wet versus dry therapeutic body wraps through an exploratory randomized controlled open label blinded outcome assessment approach.

The primary objective is the comparison of change in ABC irritability scores from baseline to 3 months between the two groups. According to the potential recruitment, we plan to recruit 30 subjects in each group. This sample size could allow us to detect a minimum effect size of 0.74 between the 2 groups (considered large in literature) with a power of 80% (two-sided test and type I error of 5%).

As described elsewhere, wet or dry session will be organized through twice-a-week sessions for a 3-month duration.

Comparison in primary outcome (ABC irritability score) between the 2 groups will be performed using Analysis of Covariance (ANCOVA) adjusted for the baseline value. The standardized difference (effect size) will be computed taking into account the adjustment for baseline and its 95% confidence interval will be estimated using a bootstrap resampling. The validity of the ANCOVA model will be checked by examining the model residuals.

The same methodology will be used for the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* a current diagnosis of autism, Asperger syndrome, atypical autism according ICD-10 criteria confirmed by specialized clinical assessment;
* presenting severe behavioural disturbances such as hetero and self-injurious behaviours, automutilation, severe motor hyperactivity, severe stereotypies.
* having a systematically consultation by a neuro pediatric.

Exclusion Criteria:

* children with known organic syndrome and/or non-stabilized neuropediatric (e.g. seizures) or medical (e.g. diabetes mellitus) comorbidities.
* patients with stabilized seizure condition, antiepileptic medication should be stable for at least 4 weeks.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist (ABC) irritability score | Baseline and 3 months
  Measure the reduction in the intensity of the behavioral disorders objectified by the sub-score Irritability of the scale ABC

SECONDARY OUTCOMES:
ABC hyperactivity score | Baseline,1-month, 2-month and 3-months
  Measure the reduction in the intensity of the behavioral disorders objectified by the sub-score hyperactivity of the scale ABC
ABC lethargy score | Baseline,1-month, 2-month and 3-months
  Measure the reduction in the intensity of the behavioral disorders objectified by the sub-score lethargy of the scale ABC
ABC inappropriate speech score | Baseline,1-month, 2-month and 3-months
  Measure the reduction in the intensity of the behavioral disorders objectified by the sub-score inappropriate speech of the scale ABC
ABC stereotypic behavior score | Baseline,1-month, 2-month and 3-months
  Measure the reduction in the intensity of the behavioral disorders objectified by the sub-score stereotypic behavior of the scale ABC
ABC Total score | Baseline,1-month, 2-month and 3-months
  Measure the reduction in the intensity of the behavioral disorders objectified by the total score of the scale ABC
Child Autism Rating Scale (CARS) | Baseline,1-month, 2-month and 3-months
  Measure the decrease in the intensity of autistic symptoms
Clinical Global Impression-Improvement (CGI-I) | Baseline,1-month, 2-month and 3-months
  Measure the global clinical outcome
Clinical Global Impression-Severity (CGI-S) | Baseline,1-month, 2-month and 3-months
  Measure the global clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Delion, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (13):
- France (13):
  - Centre de Santé Mentale Angevin, Angers
  - Centre Hospitalier d'Arras, Arras
  - Centre Hospitalier Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier Montfavet, Avignon
  - Institut Départemental Albert Calmette, Camiers
  - Centre Hospitalier de Douai, Douai
  - Etablissement Public de Santé Roger Prévot, Gennevilliers
  - Centre Hospitalier de Lens, Lens
  - Hôpital Fontan, CHRU, Lille
  - Institut Médico-éducatif, Montigny-en-Ostrevent
  - Etablissement de Santé Maison Blanche, Paris
  - Groupe Hospitalier Pitier-Salpêtrière, Paris
  - Etablissement Public de Santé Mentale Val de Lys-Artois, Saint-Venant

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Delion P, Labreuche J, Deplanque D, Cohen D, Duhamel A, Lallie C, Ravary M, Goeb JL, Medjkane F, Xavier J; Therapeutic Body Wrap Study group. Therapeutic body wraps (TBW) for treatment of severe injurious behaviour in children with autism spectrum disorder (ASD): A 3-month randomized controlled feasibility study. PLoS One. 2018 Jun 29;13(6):e0198726. doi: 10.1371/journal.pone.0198726. eCollection 2018. PMID 29958284
- [Derived] Huang HF, Tian JL, Yang XT, Sun L, Hu RY, Yan ZH, Li SS, Xie Q, Tian XB. Efficacy and safety of low-molecular-weight heparin after knee arthroscopy: A meta-analysis. PLoS One. 2018 Jun 21;13(6):e0197868. doi: 10.1371/journal.pone.0197868. eCollection 2018. PMID 29927930